CLINICAL TRIAL: NCT01176825
Title: Reducing High-Risk Behaviors Among Bipolar Patients Transitioning to Adulthood
Brief Title: Cognitive-Behavior Therapy for Young Adults With Bipolar Disorder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Aude Henin, Co-Director, Child CBT Program, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH081335 (NIH); R34MH081335 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-06 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Bipolar Disorder
Keywords: bipolar disorder; cognitive behavior therapy; alcohol abuse; drug abuse; high risk behaviors; medication adherence; psychosocial functioning
MeSH Terms: conditions — Bipolar Disorder; Alcoholism; Substance-Related Disorders; Medication Adherence | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT (Experimental): 14-week individual cognitive-behavior therapy
  Interventions: Behavioral: cognitive-behavior therapy (CBT)
- Treatment As Usual (No Intervention): 14-week waitlist control

INTERVENTIONS:
Behavioral: cognitive-behavior therapy (CBT) — 14 sessions of individual cognitive-behavior therapy. Sessions last 50-60 minutes and are held weekly. 2 optional monthly booster sessions may also be held after the end of treatment.
  Arms: CBT

SUMMARY:
The aim of the study is to develop and pilot test a cognitive-behavioral (CBT) intervention for young adults, ages 18-24 with bipolar disorder. The 14-week intervention focuses on improving management of bipolar disorder, reducing involvement in high-risk behaviors, and enhancing psychosocial functioning. The intervention also focuses on issues specific to transition-age youth. The study includes two phases: In phase 1, the intervention will be developed, refined, and openly piloted with several participants. In phase 2,the investigators will conduct a randomized clinical trial, in which 40 participants will be randomized either to receive the intervention right away, or to a 14-week waitlist condition. Participants will be evaluated at baseline, week 5, week 10, and week 14 of the study period, as well as at 3- and 6-month follow up, using measures of mood symptoms, high-risk behaviors, drug and alcohol use, and psychosocial functioning.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of bipolar spectrum disorder (Bipolar I, Bipolar II, or Bipolar NOS Disorder)
* ages 18-24 years
* able to understand the nature of the study as well as potential risks and benefits
* in treatment with a physician or nurse-practitioner for their bipolar disorder, or willing to seek and obtain such treatment if needed.

Exclusion Criteria:

* concurrent cognitive-behavioral psychotherapy
* documented mental retardation
* pervasive developmental disorder
* current serious medical illness
* inability to participate in the intervention because of acuity of symptoms
* current drug or alcohol dependence (other than marijuana dependence)

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2007-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Clinical Global Improvement Scale (CGI)-Improvement | week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Clinician-rated change in mood symptoms and overall functioning
feasibility and acceptability | post-treatment
  We will assess the percentage of completers versus drop-outs to examine feasibility of treatment procedures

SECONDARY OUTCOMES:
Adapted Y-BOCS | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  a version of the Yale-Brown Obsessive-Compulsive Scale that has been adapted to assess involvement in high-risk behaviors. This measure is individualized for each participant to assess their specific high-risk behavior that they would like to work on in treatment
Social Adjustment Scale (SAS) | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Assesses social, educational, occupational, and family functioning
Timeline Follow-Back | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Assesses alcohol and drug use over the past 30 days.
SCID depression and mania modules | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Clinician-administered measure that assesses the presence and severity of depression and mania over the past month.
Medication history and adherence | baseline, post-treatment, 6 month follow-up
  Assesses treatment with different classes of medication, psychotherapy, and psychiatric hospitalization
Adult Suicidal Ideation Questionnaire (ASIQ) | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Assesses severity of suicidal thoughts and behaviors
High-Risk Sexual Behaviors | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
Beck Hopelessness Scale | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
Barratt Impulsiveness Scale | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
Self-Control Behavior Schedule | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Assesses learned resourcefulness and self-control behaviors including problem-solving skills and self-efficacy
Hamilton Depression Scale (HAM-D) | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Clinician-administered measure that assesses severity of depressive symptoms over the past week
Young Mania Rating Scale | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
  Clinician-administered measure that assesses severity of manic symptoms over the past week.
Treatment Satisfaction Questionnaire | post-treatment
  Assesses participants' satisfaction with the treatment received
Urine Toxicology Screen | baseline, post-treatment, 6 mo follow-up
Risky Driving Inventory | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu
South Oaks Gambling Screen | baseline, week 5, week 10, week 14, 3 mo fu, 6 mo fu

CONTACTS AND LOCATIONS:
Overall Officials: Aude Henin, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States